CLINICAL TRIAL: NCT01671657
Title: US Eeva™ Pregnancy Investigational Clinical Study (US EPIC)
Acronym: US EPIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-AUX-008
Record Dates: First submitted 2012-08-21; First posted 2012-08-23 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Infertility
Keywords: In vitro fertilization; Assisted reproductive therapy; Time-lapse image recording; Image analysis software
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Eeva Test Group: Day 3 embryo transfers that used Eeva with morphology grading (Test Group).
- Matched case control group: Day 3 embryo transfers using morphology grading only (from concurrent Control Group).

SUMMARY:
The purpose of this clinical investigation is to gather data to evaluate the impact of using Eeva with traditional morphology grading on implantation rates.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to gather data to evaluate the impact of implantation rates for Day 3 embryo transfers using Eeva and morphology grading (test group) versus Day 3 embryo transfers using morphology grading only (from a concurrent control group).

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing fresh in vitro fertilization treatment using their own eggs or donor eggs.
* IVF cycle attempts ≤ 2.
* Egg age ≤ 40 years.
* Planned Day 3 embryo transfer.
* At least 4 normally fertilized eggs (2PN).
* All 2PN embryos must be imaged by Eeva.
* Ejaculated sperm or sperm from the epididymis (fresh or frozen).
* Willing to comply with study protocol and procedures.
* Willing to provide written informed consent.

Exclusion Criteria:

* Planned preimplantation genetic diagnosis or preimplantation genetic screening.
* Planned "freeze all" cycle (oocytes or embryos).
* Sperm retrieved from testicular tissue.
* Abnormal uterine cavity as evaluated by standard methods.
* Gestational carrier.
* Endometriosis
* Hydrosalpinx.
* History of cancer.
* Concurrent participation in another clinical study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing in vitro fertilization treatment who provide informed consent and plan to undergo Day 3 embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Rate of implantation | 5-6 gestational age
  To compare implantation rates for the Day 3 embryo transfers that used Eeva with morphology grading (test group) versus Day 3 embryo transfers using morphology grading only (control group).

SECONDARY OUTCOMES:
To evaluate clinical pregnancy rates from the Eeva Test group to the Control group | 5-6 weeks gestational age
Ongoing pregnancy rate | Gestational age week 8-12
Multiple pregnancy rate | Gestational age weeks 5-6 and 8-12
Spontaneous miscarriage rate | Gestational age week 8-12

CONTACTS AND LOCATIONS:
Overall Officials: Shehua Shen, MD, ELD, Study Director — Progyny, Inc.
Locations (1):
- Fertility Physicians of Northern California, San Jose, California, United States

REFERENCES:
- [Derived] Adamson GD, Abusief ME, Palao L, Witmer J, Palao LM, Gvakharia M. Improved implantation rates of day 3 embryo transfers with the use of an automated time-lapse-enabled test to aid in embryo selection. Fertil Steril. 2016 Feb;105(2):369-75.e6. doi: 10.1016/j.fertnstert.2015.10.030. Epub 2015 Nov 18. PMID 26604069